CLINICAL TRIAL: NCT06265493
Title: Postoperative Infectious Complications Calculator for Elderly Patients--A Derivation and External Validation of Prediction Models Based on Two Centers Large Sample
Brief Title: Postoperative Infectious Complications Calculator for Elderly Patients
Status: Completed | Type: Observational
Sponsor: Weidong Mi (Other)
Responsible Party: Sponsor-Investigator, Weidong Mi, Director, Department of Anesthesiology, The First Medical Center, Chinese PLA General Hospital
Organization: Chinese PLA General Hospital (Other)
Other Study IDs: PLAGH-AOC-L02
Record Dates: First submitted 2024-02-11; First posted 2024-02-20 (Actual); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Postoperative Infection; Geriatrics; Prediction
Keywords: postoperative infectious complications; elderly patients; retrospective study; prediction model; calculator

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- derivation cohort: 29785 in the derivation cohort
- internal validation cohort: 7445 in the internal validation cohort

SUMMARY:
The investigators established a first-ever convenient scoring system for clinicians to assess the risk of Postoperative infectious complications (PICs) for elderly patients. Our scoring system can aid in the early detection of potential risks for postoperative infections. Higher-score patients were more likely to experience postoperative infections.

DETAILED DESCRIPTION:
Background:

Postoperative infectious complications (PICs) are related to increased morbidity, mortality, and costs, especially in elderly patients. However, published prediction models of PICs are rarely based on elderly patients.

Objective:

The study wanted to identify practical and valuable variables that could be used to predict postoperative infections and establish a convenient scoring system for clinicians to assess the risk of such conditions in elderly patients.

Methods： Data from 2 population-based cohorts of elderly patients undergoing non-cardiac and non-neurology surgery were used to derive and validate multivariable logistic regression models. The risk prediction models were derived from 37230 patients hospitalized in the First Medical Center of the Chinese PLA General Hospital (January 2012 - August 2018). The risk prediction models were externally validated with data from a cohort of 10252 patients hospitalized in Henan Provincial People's Hospital (November 2014 to May 2022).

ELIGIBILITY:
Inclusion Criteria:

1. age ≥ 65 years and
2. patients undergoing surgery with anesthesia.

Exclusion Criteria:

1. patients undergoing neurosurgery or cardiac surgery,
2. preoperative infectious diseases, and
3. patients with ≥50% of data missing.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: A total of 37230 participants were included in the derivation and internal validation cohorts (29785 in the derivation cohort and 7445 in the internal validation cohort).
Sampling Method: Non-Probability Sample
Enrollment: 37230 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-30 (Actual)

PRIMARY OUTCOMES:
Postoperative Infectious Complications Calculator for Elderly Patients | January 2012 - August 2018
  A Derivation and External Validation of Prediction Models based on two centers large sample

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, Ph.D., Study Chair — Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital
Locations (1):
- Depatment of Anesthesiology, The First Medical Center Affiliation: Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No